CLINICAL TRIAL: NCT05988177
Title: Clinical Study on the Efficacy and Safety of Carrimycin Tablets in Hemophagocytic Lymphohistiocytosis Patients With Carbapenem-resistant Infections
Brief Title: Efficacy and Safety of Carrimycin Tablets in HLH Patients With Carbapenem-resistant Infections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Professor and Head of hematology, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH20230522002
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Carbapenem Resistant Bacterial Infection; Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — carrimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrimycin tablets (Experimental): Carrimycin tablets
  Interventions: Drug: Carrimycin tablets

INTERVENTIONS:
Drug: Carrimycin tablets — Carrimycin tablets are administered 400mg a day orally for 7 days.
  Other Names: Carrimycin

SUMMARY:
This study aimed to investigate the efficacy and safety of Carrimycin tablets in hemophagocytic lymphohistiocytosis patients with Carbapenem-resistant infections.

DETAILED DESCRIPTION:
Hemophagocytic lymphohistiocytosis (HLH) is a critical condition characterized by the undue activation of cytotoxic T lymphocytes, natural killer cells, and macrophages, resulting in excessive secretion of infammatory cytokines. Infection is an important trigger for HLH. This study aimed to investigate the efficacy and safety of Carrimycin tablets in hemophagocytic lymphohistiocytosis patients with Carbapenem-resistant infections.

ELIGIBILITY:
Inclusion Criteria:

* Met HLH-2004 diagnostic criteria;
* Active infection；
* Empirical treatment with carbapenems did not respond after 72 hours；
* Age >18 years old, no gender limitation;
* Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

* Other antibiotics should be selected according to the results of drug sensitivity；
* Systemic antibiotics other than carbapenems are used with 72 hours；
* Inability to take oral medications due to disease of gastrointestinal tract；
* Severe liver insufficiency;
* Expected survival time < 1 month;
* Pregnant or breasting-feeding women;
* Allergic to Carrimycin tablets;
* Active hepatitis B or hepatitis C infection;
* Patients with HIV infection;
* Patients with other contraindications considered unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cure rates of infections | 1 week and 2 weeks after initiation of treatment
  The percentage of participants having clinical cure
Overall response rate of HLH | 2 weeks after treatment
  Overall response rate includes complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
Overall Survival | 1 years
  OS will be assessed from initiation of treatment to death from any cause
Incidence and Severity of Adverse Events | 28 days
  Treatment-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No